CLINICAL TRIAL: NCT06833684
Title: Intermittent Colonic Exoperistalsis Treatment With MOWOOT Medical Device to Treat Chronic Constipation in Adult Patients Waiting for Using Trans-Anal Irrigation: A Pilot Study
Brief Title: MowOot and Trans-anal Irrigation fOr coNstipation
Acronym: MOTION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: usMIMA S.L. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOW-08-2024
Record Dates: First submitted 2025-02-12; First posted 2025-02-19 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Constipation Chronic Idiopathic
Keywords: constipation; transit problems; Trans-Anal Irrigation; Intermittent Colonic Exoperistalsis
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: This is a prospective, open-labelled, longitudinal, controlled study, with two treatment groups, performed at one single centre. For both groups, patients will be their own control in the pre and post analysis of primary and secondary outcomes.
Masking Description: This is an open-label study, meaning there is no masking. Both the participants and the researchers are aware of the treatment being administered. This approach is necessary due to the nature of the intervention, which makes blinding impractical.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental ICE Group (Experimental): Each patient will receive 1 ICE treatment of 20 minutes at least once per day, every day at the same hour, during the intervention period of 12 weeks.
  Interventions: Device: ICE Treatment
- Control TAI Group (Active Comparator): Each patient will follow the usual TAI standard-of-care treatment for the intervention period of 12 weeks.
  Interventions: Procedure: TAI Standard-of-Care Treatment

INTERVENTIONS:
Device: ICE Treatment — Each patient in the Experimental ICE Group will receive one Intermittent Colonic Exoperistalsis (ICE) treatment session lasting 20 minutes. These sessions will be conducted at least once per day, every day at the same hour, for a total duration of 12 weeks. The ICE treatment involves using the MOWOOT medical device designed to alleviate chronic constipation by stimulating colonic peristalsis.
  Arms: Experimental ICE Group
Procedure: TAI Standard-of-Care Treatment — Each patient in the Control TAI Group will follow the usual Trans-Anal Irrigation (TAI) standard-of-care treatment. This involves the regular use of TAI procedures as prescribed by healthcare professionals for the intervention period of 12 weeks. The TAI treatment is a well-established method for managing chronic constipation by mechanically clearing the bowel.
  Arms: Control TAI Group

SUMMARY:
This prospective, open-labelled, longitudinal, controlled study aims to evaluate the suitability of Intermittent Colonic Exoperistalsis (ICE) treatment for adults with refractory chronic constipation who are awaiting trans-anal irrigation (TAI). The ICE treatment will be applied using the MOWOOT device (USMIMA). The study involves two treatment groups: an experimental group receiving daily ICE treatments and a control group following standard TAI care. Participants will serve as their own controls in pre- and post-treatment analyses to assess changes in bowel management satisfaction and other outcomes.

DETAILED DESCRIPTION:
This study is a prospective, open-labelled, longitudinal, controlled trial conducted at a single center. It aims to assess the suitability of Intermittent Colonic Exoperistalsis (ICE) treatment for bowel management in adults with refractory chronic constipation who are awaiting trans-anal irrigation (TAI). The ICE treatment will be applied using the MOWOOT device (USMIMA). The study includes two treatment groups:

Experimental ICE Group: Participants will receive one ICE treatment session lasting 20 minutes daily, at the same hour, for 12 weeks.

Control TAI Group: Participants will follow the usual TAI standard-of-care treatment for 12 weeks.

Participants will be given the option to choose between the ICE treatment and the TAI treatment after both options are explained to them. Healthcare professionals will recommend the most suitable treatment based on individual patient needs, but the final decision will rest with the patients.

The primary objective is to evaluate the change in satisfaction with daily quality of life related to bowel management, measured by a Likert scale (Bothersome scale). Secondary objectives include assessing the efficacy of the ICE treatment on chronic constipation, both qualitatively and quantitatively, and evaluating the economic impact from the hospital's perspective.

Secondary outcomes will be measured through various patient-reported and health professional-reported metrics, including changes in quality of life (PAC-QOL), constipation symptoms (PAC-SYM), constipation severity (CCCS), time spent in bowel management and evacuation, use of other treatments, number of consultations and hospital admissions, productivity, acceptability and ease of use of the ICE treatment, reported problems, compliance, adherence, and persistence in treatment. Health professional outcomes will include time spent per visit, total time spent until independent use of MOWOOT, ease of patient management, and patient treatment preferences.

ELIGIBILITY:
Inclusion Criteria:

1. Adult people (18 yo or older) of any gender
2. Attending their pre-scheduled on-site visit to the site (The Sir Alan Parks Physiology & Pelvic Floor Biofeedback Unit | Central Middlesex Hospital) due to constipation (Symptoms meeting the American College of Gastroenterology definition of chronic constipation: unsatisfactory defaecation characterized by infrequent stool, difficult stool passage or both for at least previous 3 months.
3. Bothered by their constipation
4. Failed biofeedback (in absence of outlet problems)
5. In waiting list to use TAI
6. Able to undertake the treatment with the MOWOOT device or TAI themselves, or with a carer willing to do it
7. Able to understand the study requirements
8. Able to understand written and spoken English (due to questionnaire validity)
9. Able and willing to provide written informed consent to participate

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

Disease phenotype exclusion criteria:

* Irritable Bowel Syndrome with Diarrhoea (IBS-D) or alternating constipation and diarrhoea (IBSmix): (not due to laxative use)
* Inflammatory Bowel Disease (IBD)
* Significant outlet problem
* Trapping rectocele
* Intra anal rectal intussusception
* External rectal prolapse

Device-related exclusion criteria:

* Abdominal perimeter ≤65cm or ≥130cm
* Unable to independently use the MOWOOT technology, unless a carer is available daily to assist

Other medical conditions, medications and contraindications:

* Pregnancy or attempt to become pregnant in the next 6 months.
* Previous large bowel resection
* Active anorexia or bulimia
* Active abdominal cancer
* Large inguinal or umbilical hernia
* Recent abdominal scars, abdominal wounds or skin disorders that may make abdominal massage uncomfortable
* Any condition that contraindicates abdominal massage.
* Significant abdominal pain
* Participation in another parallel interventional clinical trial or less than 2 months from participation in a previous interventional clinical trial
* Planned surgery* if it might be within trial dates (* minor surgery not affecting adherence to treatment is allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Satisfaction with Daily Quality of Life Related to Bowel Management | 12 weeks
  Assessed by the Bothersome Scale (a Likert scale) where 0 is 'not at all' and 10 is 'a great deal,' with higher scores indicating a worse outcome

SECONDARY OUTCOMES:
Changes in Quality of Life According to PAC-QOL Score | 12 weeks
  Assessed by the PAC-QOL (Patient Assessment of Constipation Quality of Life) scale, where higher scores indicate a worse quality of life.
Changes in Constipation Symptoms According to PAC-SYM Score | 12 weeks
  Measured using the PAC-SYM (Patient Assessment of Constipation Symptoms) scale, with higher scores reflecting more severe constipation symptoms
Changes in Constipation Severity According to CCCS | 12 weeks
  Evaluated by the CCCS (Constipation Clinical Severity Scale), where higher scores denote greater severity of constipation
Change in Time Spent in Bowel Management | 12 weeks
  Measured in minutes per day, data from bowel diaries.
Change in Time Spent in Evacuation | 12 weeks
  Measured in minutes per day, data from bowel diaries.
Change in Use of Other Treatments (e.g., Laxatives, Suppositories) | 12 weeks
  Data from patient surveys.
Change in Number of Consultations to Primary Care (GP, Nurse) | 12 weeks
  Data from patient surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Thomas, MD, PhD, Principal Investigator — The Sir Alan Parks Physiology & Pelvic Floor Biofeedback Unit | Central Middlesex Hospital
Locations (1):
- The Sir Alan Parks Physiology & Pelvic Floor Biofeedback Unit., Central Hospital, Department of Physiology, St Mark's Hospital, The National Bowel Hospital, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No